CLINICAL TRIAL: NCT07327385
Title: The Pathophysiological Mechanisms and Novel Treatments Linking Stress and Mental Health Conditions -To Investigate the Change of Brain and Autonomic Function From Different Protocols of Repeated Transcranial Magnetic Stimulation Therapy for Patients With Post-traumatic Stress Disorder Comorbid Major Depressive Disorder: a Randomized, Double-blind, Crossover Study.
Brief Title: To Investigate the Change of Brain and Autonomic Function From Different Protocols of Repeated Transcranial Magnetic Stimulation Therapy for Patients With Post-traumatic Stress Disorder Comorbid Major Depressive Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Tien-Yu Chen, Visiting Physician, Tri-Service General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C202405067
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Posttraumatic Stress Disorder (PTSD); Depression - Major Depressive Disorder
Keywords: PTSD; functional near-infrared spectroscopy; Heart Rate Variability; HRV; rTMS
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, double-blind, sham-controlled, crossover design to examine the immediate neurophysiological effects of noninvasive brain stimulation in patients with posttraumatic stress disorder comorbid with major depressive disorder. Each participant receives both an active stimulation session (either prolonged intermittent theta-burst stimulation or high-frequency repetitive transcranial magnetic stimulation) and a sham stimulation session in a randomized sequence. A washout period of 7 days is implemented between sessions to minimize potential carryover effects. Blinding is maintained for participants and outcome assessors, while stimulation operators are not involved in outcome evaluation. Prefrontal cortical activity and autonomic nervous system responses are assessed immediately before and after each stimulation session.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will be blinded to treatment assignment. Active and sham stimulation will be delivered using coils identical in appearance and sound. The stimulation operator will not participate in clinical or physiological outcome assessments. Blinding codes will remain concealed until completion of data collection and database lock.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged iTBS With Sham Control (Experimental): Participants in this arm receive a single-session prolonged intermittent theta-burst stimulation (prolonged iTBS) targeting the right dorsolateral prefrontal cortex, as well as a sham stimulation session in a randomized crossover sequence. Each stimulation session is separated by a 7-day washout period. Neurophysiological and autonomic measures are obtained immediately before and after each session.
  Interventions: Device: Prolonged Intermittent Theta-Burst Stimulation (prolonged iTBS); Device: Sham Transcranial Magnetic Stimulation
- HF-rTMS With Sham Control (Experimental): Participants in this arm receive a single-session high-frequency repetitive transcranial magnetic stimulation (HF-rTMS) targeting the right dorsolateral prefrontal cortex, as well as a sham stimulation session in a randomized crossover sequence. Each stimulation session is separated by a 7-day washout period. Neurophysiological and autonomic measures are obtained immediately before and after each session.
  Interventions: Device: High-Frequency Repetitive Transcranial Magnetic Stimulation (HF-rTMS); Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Prolonged Intermittent Theta-Burst Stimulation (prolonged iTBS) — Prolonged intermittent theta-burst stimulation is delivered using a Magstim Rapid2 stimulator with a figure-eight coil targeting the right dorsolateral prefrontal cortex (DLPFC), localized with the Beam F4 method. Stimulation is administered at 80% of individual motor threshold using an intermittent theta-burst pattern (2 seconds on, 8 seconds off), consisting of 3-pulse bursts at 50 Hz repeated at 5 Hz. A single session lasts approximately 9.5 minutes and delivers a total of 1,800 pulses.
  Arms: Prolonged iTBS With Sham Control
Device: High-Frequency Repetitive Transcranial Magnetic Stimulation (HF-rTMS) — High-frequency rTMS is delivered using a Magstim Rapid2 stimulator with a figure-eight coil targeting the right dorsolateral prefrontal cortex (DLPFC), localized with the Beam F4 method. Stimulation follows the DASH protocol at 120% of motor threshold and 10 Hz frequency, with 4-second stimulation trains (40 pulses per train) followed by an 11-second inter-train interval, for a total of 75 trains. The single-session duration is approximately 18.75 minutes, delivering 3,000 pulses.
  Arms: HF-rTMS With Sham Control
Device: Sham Transcranial Magnetic Stimulation — Sham stimulation is delivered using a placebo coil identical in appearance and acoustic output to the active coil but without producing a magnetic field sufficient to induce cortical stimulation. Sham sessions match the corresponding active stimulation protocol in duration and procedure to maintain blinding.

SUMMARY:
This study aims to investigate the immediate neurophysiological and autonomic effects of two noninvasive brain stimulation protocols-prolonged intermittent theta-burst stimulation (prolonged iTBS) and high-frequency repetitive transcranial magnetic stimulation (HF-rTMS)-in patients with posttraumatic stress disorder (PTSD) comorbid with major depressive disorder (MDD). Using a randomized, double-blind, sham-controlled crossover design, changes in prefrontal cortical activity measured by functional near-infrared spectroscopy (fNIRS) and autonomic nervous system function measured by heart rate variability (HRV) will be assessed before and immediately after a single stimulation session.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a chronic psychiatric condition frequently accompanied by depressive symptoms and autonomic dysregulation. Although pharmacotherapy and psychotherapy are standard treatments, many patients show limited response or experience significant side effects. Repetitive transcranial magnetic stimulation (rTMS) has emerged as a promising noninvasive neuromodulatory intervention; however, the optimal stimulation protocol for PTSD remains unclear.

This randomized, double-blind, crossover study is designed to compare the immediate effects of prolonged iTBS and HF-rTMS applied to the right dorsolateral prefrontal cortex (DLPFC) on brain function and autonomic regulation in adults with PTSD comorbid with MDD. Each participant will receive one active stimulation session (either prolonged iTBS or HF-rTMS) and one sham stimulation session in a randomized order, separated by a 7-day washout period to minimize carryover effects.

Prefrontal cortical activation will be measured using multi-channel functional near-infrared spectroscopy (fNIRS), and autonomic nervous system activity will be assessed using heart rate variability (HRV) analysis derived from electrocardiographic recordings. The primary objective is to characterize protocol-specific neurophysiological response patterns and identify quantifiable biomarkers of brain stimulation response that may inform future personalized treatment strategies for PTSD with comorbid depression.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 65 years.
2. Clinical diagnosis of posttraumatic stress disorder (PTSD) according to DSM-5 criteria, confirmed by a board-certified psychiatrist.
3. Presence of comorbid major depressive disorder with stable clinical condition.
4. PTSD symptom severity defined as: PTSD Checklist for DSM-5, Chinese version (C-PCL-5) total score ≥ 31.
5. Depressive symptom severity defined as: Patient Health Questionnaire-9 (PHQ-9) total score ≥ 10.
6. Stable psychiatric medication regimen for at least 4 weeks prior to enrollment, or medication-free.
7. Ability to understand the study procedures and provide written informed consent.
8. Normal or corrected-to-normal vision and hearing.
9. Ability to comply with study procedures and visit schedule.

Exclusion Criteria:

1. Lifetime diagnosis of schizophrenia spectrum disorders, bipolar disorder, or pervasive developmental disorders.
2. Alcohol or substance use disorder (excluding caffeine and nicotine) within the past 6 months.
3. Ongoing trauma-focused psychotherapy during the study period.
4. Prior exposure to repetitive TMS treatment exceeding five sessions.
5. Current or recent (within the past year) suicidal ideation or behavior, defined as: PHQ-9 item 9 score ≥ 1, confirmed by clinical psychiatric evaluation.
6. Self-injurious behavior requiring medical attention within the past 3 months.
7. History of epilepsy, seizure disorder, or family history of epilepsy.
8. Significant neurological disorders, severe traumatic brain injury, or history of brain surgery.
9. Presence of implanted metallic or electronic medical devices (e.g., pacemakers, cochlear implants, neurostimulators).
10. Uncontrolled major medical illnesses or severe cardiovascular disease.
11. Pregnancy or breastfeeding.
12. Skin lesions or infections at the stimulation site.
13. Use of medications known to significantly lower seizure threshold (e.g., tricyclic antidepressants or certain analgesics).
14. Any condition deemed by the investigator to render the participant unsuitable for rTMS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-17 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Prefrontal Cortical Activation | Immediately before stimulation and immediately after each single stimulation session (active and sham), within each study period
  Change in prefrontal cortical activation, measured as differences in oxygenated hemoglobin (HbO₂) concentration using multi-channel functional near-infrared spectroscopy (fNIRS). Measurements are obtained at rest immediately before and immediately after each stimulation session to assess acute neurophysiological effects of prolonged intermittent theta-burst stimulation and high-frequency repetitive transcranial magnetic stimulation.

SECONDARY OUTCOMES:
Change in Autonomic Nervous System Activity | Immediately before stimulation and immediately after each single stimulation session (active and sham), within each study period
  Autonomic nervous system activity assessed by heart rate variability (HRV) derived from 5-minute resting-state electrocardiographic recordings. HRV parameters are analyzed to evaluate acute changes in autonomic regulation following active versus sham brain stimulation.
Incidence of Adverse Events | From the start of the first stimulation session through 7 days after the second stimulation session
  Frequency and type of adverse events, including local discomfort, headache, dizziness, autonomic symptoms, or other reported events, assessed using standardized safety checklists immediately after stimulation, during 24-hour follow-up, and at post-study visit.
Change in PTSD Symptom Severity | Baseline, before the second stimulation session (Day 8), and 7 days after completion of the crossover phase
  Change in posttraumatic stress disorder symptom severity measured by the PTSD Checklist for DSM-5, Chinese version (C-PCL-5), used to monitor symptom stability and safety during the crossover study.
Change in Depressive Symptom Severity | Baseline, before the second stimulation session (Day 8), and 7 days after completion of the crossover phase
  Change in depressive symptom severity assessed using the Patient Health Questionnaire-9 (PHQ-9), primarily for safety monitoring and detection of symptom exacerbation during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Tien-Yu Chen, PhD, MD, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Neihu, Taiwan